CLINICAL TRIAL: NCT01220622
Title: Nimodipine Preventing Cognitive Impairment in Ischemic Cerebrovascular Events: A Randomized, Placebo-Controlled, Double-Blind Trial (NICE)
Brief Title: Efficacy and Safety Study of Nimodipine to Prevent Mild Cognitive Impairment After Acute Ischemic Strokes
Acronym: NICE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Yongjun Wang, Beijing Tian Tan Hospital, Capital Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BSP-SOP-040
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Stroke; Mild Cognitive Impairment
Keywords: Stroke; Mild cognitive impairment; Nimodipine
MeSH Terms: conditions — Stroke; Cognitive Dysfunction | interventions — Nimodipine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nimodipine (Active Comparator)
  Interventions: Drug: Nimodipine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nimodipine — Administration of nimodipine 30mg tid for 6 months
  Other Names: Nimodiping Pian
  Arms: Nimodipine
Drug: Placebo — Administration of placebo 30mg tid for 6 months
  Other Names: Control group
  Arms: Placebo

SUMMARY:
The trial was designed to test the hypothesis that early treatment with nimodipine has a positive effect on cognition impairment after acute ischemic stroke.

DETAILED DESCRIPTION:
656 patients diagnosed with acute cerebral ischemia disease (onset≤7d) based on ICD-10 and CT/MRI criteria, who have cognitive impairment meeting all of the inclusion criteria and none of the exclusion criteria, will be included and randomized into nimodipine treatment group and the controlled group.Evaluations of cognitive function will be taken at baseline, 1 month, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects between 30 and 80 years.
* 2. ICD-10 and CT/MRI criteria for acute cerebral infarction.
* 3. Stroke within 7 days after onset.
* 4.based on years of education correction.MMSE>17(illiteracy),MMSE>20(primary school),MMSE>24(others)
* 5. MoCA≤26 at baseline.
* 6.Hachinski ischemic score ≥7 at baseline.
* 7.Expected good compliance to study.
* 8.Informed consent signed.

Exclusion Criteria:

* 1.Diagnosis of schizophrenia, major anxiety syndrome, major depression.
* 2.Alzheimer disease, Parkinson disease, Huntington disease, and fronto-temporal dementia.
* 3.Dementia caused by (e.g., central nervous system trauma, tumor, infections, metabolic disorders, normal pressure hydrocephalus, lack of folic acid or vitamin B12, or thyroid hormone deficiency).
* 4.Contraindications to dihydropyridine derivatives.
* 5.Aphasia or other diseases that affect cognitive evaluation.
* 6.Serious arrhythmias, bradycardia (<50 bpm) or tachycardia (>120 bpm); myocardial infarction within the past 6 months; blood pressure <90/60mmHg; severe renal or hepatic insufficiency; severe anemia, Hb<100g/L; severe gastrointestinal disorders; tumor.
* 7.History of epilepsy, use of the antiepileptic drugs.
* 8.CT/MRI showed neurodegenerative changes or other lesions except cerebral ischemia.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-04 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of nimodipine on the cognitive function after acute cerebral ischemia with ADAS-cog and MMSE at 6 months in the ITT population | 6 months

SECONDARY OUTCOMES:
Assess the effect of nimodipine on the cognitive function after acute cerebral ischemia with MoCA and FAB at 6 months in the ITT population | 6 months
The prevalence of possible vascular dementia diagnosed by NINDS-AIREN criteria at 6 months | 6 months
Assess the effect of nimodipine on the cognitive function after acute cerebral ischemia with ADAS-cog and MMSE at 3 months in the ITT population | 3 months
Assess the effect of nimodipine on the cognitive function after acute cerebral ischemia with MoCA and FAB at 3 months in the ITT population | 3 months
The prevalence of possible vascular dementia diagnosed by NINDS-AIREN criteria at 1 month | 1 month
The prevalence of possible vascular dementia diagnosed by NINDS-AIREN criteria at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Wang Yongjun, M.D., Principal Investigator — Beijing Tian Tan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tian Tan Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Zheng H, Wang Y, Wang A, Li H, Wang D, Zhao X, Wang P, Shen H, Zuo L, Pan Y, Li Z, Meng X, Wang X, Shi W, Ju Y, Liu L, Dong K, Wang C, Sui R, Xue R, Pan X, Niu X, Luo B, Sui Y, Wang H, Feng T, Wang Y; NICE trial group. The efficacy and safety of nimodipine in acute ischemic stroke patients with mild cognitive impairment: a double-blind, randomized, placebo-controlled trial. Sci Bull (Beijing). 2019 Jan 30;64(2):101-107. doi: 10.1016/j.scib.2018.12.006. Epub 2018 Dec 8. PMID 36659633